CLINICAL TRIAL: NCT03058575
Title: A Randomized, Controlled, Crossover Study to Evaluate the Effects of a Novel Food Product Containing Microbiota Accessible Carbohydrates on the Human Microbiome and Associated Parameters
Brief Title: Effects of a Novel Food Product Containing Microbiota Accessible Carbohydrates on the Human Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Access Business Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BIO-1611
Record Dates: First submitted 2017-01-24; First posted 2017-02-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Gut Microbiome
Keywords: Microbiome; Gut; Skin; Fiber; Starch

STUDY DESIGN:
Intervention Model Description: This is a randomized, 2-period crossover study.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessors will be blind to who is on Arm1 and who is on Arm 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary MACs (Experimental): Dietary fiber supplement (blend of resistant starch and dietary fiber food ingredients providing 15g of microbiota accessible carbohydrate/1 scoop serving) will be provided in a powder that will be mixed with 6-10 oz of water (depending on desired thickness) and consumed as a chocolate shake.
  Interventions: Dietary Supplement: Dietary MACs
- Control (Other): No Intervention
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Dietary MACs — All subjects will have a dose-escalation period when randomized to the active arm that will occur as follows:
  Day 1: 1 scoop of product (morning, in the clinic)
  Day 2: 1 scoop of product (morning)
  Day 3: 2 scoops of product (morning and evening)
  Day 4: 2 scoops of product (morning and evening)
  Days 5-60: 3 scoops of product (morning, afternoon, evening)
  Other Names:
  Dietary fiber supplement
  Arms: Dietary MACs
Other: Control — No Intervention for 8 weeks
  Arms: Control

SUMMARY:
This is a randomized, 2-period crossover study aimed at assessing the effect of taking a food supplement containing a blend of microbial accessible carbohydrates on the diversity of the gut microbiome. Impacts to the skin, scalp and oral microbiomes; blood inflammatory biomarkers; quality and quantity of sleep; gastrointestinal quality of life; bowel habits, and facial skin features will also be evaluated.

DETAILED DESCRIPTION:
The human body is home to trillions of microbes, which have been shown to play important roles in many aspects of human biology, such as immune function and metabolism. Research in this area has primarily focused on the role that dietary factors have in modulating the gastrointestinal (GI) microbiota with associated changes in host health parameters. Specifically, dietary microbiota accessible carbohydrates (MACs), which include compounds such as resistant starches and other dietary fibers that are typically resistant to digestion, have been shown to serve as a primary source of energy for the distal gut microbiota. Metabolism of MACs by the GI microbiota is important in shaping this microbial ecosystem. A Western diet, typically low in MAC content (e.g., dietary fiber), is associated with a marked reduction in microbial diversity and depletion of specific types of potentially beneficial microbes.

Until only recently, the bulk of microbiota studies have been conducted in animals, and human studies on the GI microbiota have focused primarily on delineating the gut bacterial composition and corresponding changes in taxonomy in response to a particular dietary intervention (e.g., with prebiotics). Additionally, investigations on dietary factors influencing the skin (or scalp) and oral cavity microbiomes have only recently garnered attention. Human intervention studies that increase consumption of dietary MACs are needed to better understand how changes in the composition and function of these bacteria influence host parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 40-60 years of age, inclusive.
* Subject has a waist circumference ≥102 cm (40 inches) in men or ≥89 cm (35 inches) in women at visit 1a (week -1).
* Subject does not smoke or use any products containing nicotine (including use of any tobacco products) for the past 6 months prior to Visit 1b and has no plans to change smoking habits during the study period.
* For males, subject is willing to shave prior to facial imaging test days (total of 6 clinic visits).
* Subject is willing and able to comply with the visit schedule and fecal sample collection requirements (a total of 8 fecal samples) during the study period.
* Subject does not plan to willingly change his or her habitual diet, physical activity patterns, or body weight during the study period.
* Subject is willing and able to consume a low-calorie, 6-10 oz chocolate shake, as directed, for 8 weeks.
* Subject has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the Investigator on the basis of medical history and routine laboratory test results.
* Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

* Subject has abnormal laboratory test results of clinical significance at Visit 1b (week -1), at the discretion of the Investigator. One re-test will be allowed on a separate day prior to Visit 2 (week 0), for subjects with abnormal laboratory test results.
* Subject has a history or presence of clinically important endocrine (including hyperparathyroidism, type 1 or 2 diabetes mellitus and/or hypoglycemia), cardiovascular (including, but not limited to history of myocardial infarction, peripheral arterial disease, stroke), pulmonary (including uncontrolled asthma), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, rheumatic (including gout), biliary, and/or psychiatric disorders, that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
* Subject has had a recent (within 2 weeks of Visit 1b; week -1) episode of acute GI illness such as nausea/vomiting or diarrhea.
* Subject has a history or presence of a diagnosed GI disease, including but not limited to, irritable bowel syndrome, inflammatory bowel disease, Celiac disease, or Crohn's disease.
* Subject has a recent history (within 6 weeks of Visit 1b, week -1) of constipation (defined as <3 bowel movements per week).
* Subject has a history or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Subject has a history of bariatric surgery for weight reducing purposes.
* Subject has extreme dietary habits, including but not limited to, intentional consumption of a high fiber diet, and/or vegan/other vegetarian diets, in the opinion of the Investigator.
* Subject has had a weight loss or gain >4.5 kg in the 6 months prior to Visit 1b (week -1).
* Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) as defined by the blood pressure measured at Visit 1b (week -1). One re-test will be allowed on a separate day prior to Visit 2 (week 0), for subjects whose blood pressure exceeds either of these cut points, in the judgment of the Investigator.
* Subject has used any antibiotics within 3 months of Visit 2 (week 0).
* Subject has used medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to prebiotics or probiotics, laxatives, enemas, fiber supplements, suppositories, anti-diarrheal agents, and/or anti-spasmodics within 2 weeks of Visit 2 (week 0).
* Subject uses non-steroidal, anti-inflammatory drugs on a daily basis.
* Subject uses antacids, proton pump inhibitors, or histamine blockers on a daily basis within 1 week of Visit 2 (week 0).
* Subject has started lipid lowering prescription medication(s) within 4 weeks of Visit 2 (week 0). Subjects must be on a stable dose (defined as consistent dose) for at least 4 weeks prior to Visit 2 (week 0) and throughout the study period.
* Subject has a known allergy or sensitivity to any component or ingredient in the study product.
* Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period. The method of contraception must be recorded in the source documentation.
* Subject is a premenopausal female using a form of contraception that does not result in a normal menstrual cycle (normal cycle defined as a 21 to 35 d).
* Subject has a recent history of (within 1 month of Visit 1b) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week or more than 4 drinks at any one time (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
* Subject has been exposed to any non-registered drug product within 30 d prior to Visit 1b (week -1).
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Fecal Microbiome Shannon Diversity Index | Baseline, 2, 4 and 8 Weeks
  The Shannon Diversity Index of the fecal microbiome will be measured at each of the time points via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing

SECONDARY OUTCOMES:
Change from Baseline in Fecal Microbiome Composition | Baseline, 2, 4 and 8 Weeks
  The fecal microbial composition will be measured via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing
Change from Baseline in Forehead Skin Microbiome Composition | Baseline, 2, 4 and 8 Weeks
  The forehead skin microbial composition will be measured via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing
Change from Baseline in Scalp Skin Microbiome Composition | Baseline, 2, 4 and 8 Weeks
  The scalp skin microbial composition will be measured via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing
Change from Baseline in Oral (Buccal) Microbiome Composition | Baseline, 2, 4 and 8 Weeks
  The oral microbial composition will be measured via taxonomic profiling using 16S ribosomal RNA gene amplicon sequencing
Change from Baseline in Fecal Short Chain Fatty Acids (Butyrate) | Baseline, 2, 4 and 8 Weeks
  Fecal short chain fatty acids (e.g., butyrate) will be measured at each of the time points.
Change from Baseline in Blood Inflammatory Marker (C-Reactive Protein) | Baseline, 4 and 8 Weeks
  The inflammatory marker C-Reactive Protein in the blood will be measured at each of the time points.
Change from Baseline in Blood Inflammatory Marker (IL-10) | Baseline, 4 and 8 Weeks
  The inflammatory marker IL-10 in the blood will be measured at each of the time points.
Change from Baseline in Blood Inflammatory Marker (IL-6) | Baseline, 4 and 8 Weeks
  The inflammation marker IL-6 in the blood will be measured at each of the time points.
Change from Baseline in Blood Inflammatory Marker (TNF-Alpha) | Baseline, 4 and 8 Weeks
  The inflammation marker TNF-alpha in the blood will be measured at each of the time points.
Change from Baseline in Blood Inflammatory Marker (Lipopolysaccharides) | Baseline, 4 and 8 Weeks
  The inflammation marker lipopolysaccharides in the blood will be measured at each of the time points.
Change from Baseline in Blood Testosterone Hormone Levels | Baseline and 8 Weeks
  Blood Testosterone Levels (free and total) will be measured at each of the time points.
Change from Baseline in Blood Estradiol Levels | Baseline and 8 Weeks
  Blood Estradiol Levels will be measured at each of the time points
Change from Baseline in Fasting Blood Lipid Profiles | Baseline and 8 Weeks
  Blood lipid profiles (including total cholesterol, HDL-cholesterol, non-HDL-cholesterol, calculated LDL-cholesterol, and triglycerides) will be measured at each of the time points
Change from Baseline in Satiety | Baseline, 2, 4 and 8 Weeks
  An appetite questionnaire will be used to measure satiety at each of the time points
Change from Baseline in Heart Rate Variance | Baseline, 4 and 8 Weeks
  Heart Rate Variance will be measured using a standardized method at each of the time points
Change from Baseline in Bowel habits | Baseline, 2, 4 and 8 weeks
  Bowel habits will be recorded using a diary at each of the time points.
Change from Baseline in Stool Quality | Baseline, 2, 4 and 8 Weeks
  Subjects will record the quality of their stool using the Bristol Stool Scale at each of the time points
Change in Gastrointestinal Quality of Life (GIQOL) | 4 and 8 Weeks
  The electronic GIQOL Instrument will be used to asses GI QoL at each of the time points.
Change in Sleep Quantity | Baseline through 8 Weeks
  Each subject will wear an activity tracker (Actigraph) to measure the amount of sleep obtained from baseline to 8 weeks.
Change from Baseline in Sleep Quality | Baseline, 4 and 8 Weeks
  The electronic Pittsburgh Sleep Quality Index Instrument will be used to measure the change from baseline in Sleep Quality Index
Change from Baseline in Facial Wrinkling | Baseline, 4 and 8 Weeks
  Standardized facial images will be captured using the VISIA CR facial imaging system under multiple lighting modalities. Images will be analyzed using quantitative image analysis to assess facial wrinkling around the eye (crow's feet wrinkles).
Change from Baseline in Facial Hyperpigmentation | Baseline, 4 and 8 Weeks
  Standardized facial images will be captured using the VISIA CR facial imaging system under multiple lighting modalities. Images will be analyzed using quantitative image analysis to assess facial hyperpigmentation around the eyes and on the left and right cheeks.
Change from Baseline in Facial Redness | Baseline, 4 and 8 Weeks
  Standardized facial images will be captured using the VISIA CR facial imaging system under multiple lighting modalities. Images will be analyzed using quantitative image analysis to assess facial red features on the left and right cheeks.
Change from Baseline in Facial Porphyrins | Baseline, 4 and 8 Weeks
  Standardized facial images will be captured using the VISIA CR facial imaging system under multiple lighting modalities. Images will be analyzed using quantitative image analysis to assess facial porphyrins on the forehead, nose and on the left and right cheeks.
Change from Baseline in Facial Skin Texture | Baseline, 4 and 8 Weeks
  Standardized facial images will be captured using the VISIA CR facial imaging system under multiple lighting modalities. Images will be analyzed using quantitative image analysis to assess facial skin texture on the left and right cheeks.
Change from Baseline in Facial Skin Pores | Baseline, 4 and 8 Weeks
  Standardized facial images will be captured using the VISIA CR facial imaging system under multiple lighting modalities. Images will be analyzed using quantitative image analysis to assess facial skin pores on the left and right cheeks.
Beauty Quality of Life | 8 Weeks
  The electronic Beauty Quality of Life Instrument will be used to measure BeautyQOL at 8 Weeks
Test Product Likability | 8 Weeks
  An electronic product likability questionnaire will be used to measure the subjects response to how much they liked the test product at 8 weeks. Product attributes will include flavor, sweetness, texture, thickness, and ease of consumption.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Lawless, MD, Principal Investigator — Biofortis Innovation Research
Locations (1):
- Biofortis Innovation Services, Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beresniak A, de Linares Y, Krueger GG, Talarico S, Tsutani K, Duru G, Berger G. Validation of a new international quality-of-life instrument specific to cosmetics and physical appearance: BeautyQoL questionnaire. Arch Dermatol. 2012 Nov;148(11):1275-82. doi: 10.1001/archdermatol.2012.2696. PMID 23165832
- [Background] De Filippo C, Cavalieri D, Di Paola M, Ramazzotti M, Poullet JB, Massart S, Collini S, Pieraccini G, Lionetti P. Impact of diet in shaping gut microbiota revealed by a comparative study in children from Europe and rural Africa. Proc Natl Acad Sci U S A. 2010 Aug 17;107(33):14691-6. doi: 10.1073/pnas.1005963107. Epub 2010 Aug 2. PMID 20679230
- [Background] El Kaoutari A, Armougom F, Gordon JI, Raoult D, Henrissat B. The abundance and variety of carbohydrate-active enzymes in the human gut microbiota. Nat Rev Microbiol. 2013 Jul;11(7):497-504. doi: 10.1038/nrmicro3050. Epub 2013 Jun 10. PMID 23748339
- [Background] Eypasch E, Williams JI, Wood-Dauphinee S, Ure BM, Schmulling C, Neugebauer E, Troidl H. Gastrointestinal Quality of Life Index: development, validation and application of a new instrument. Br J Surg. 1995 Feb;82(2):216-22. doi: 10.1002/bjs.1800820229. PMID 7749697
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] Karlsson F, Tremaroli V, Nielsen J, Backhed F. Assessing the human gut microbiota in metabolic diseases. Diabetes. 2013 Oct;62(10):3341-9. doi: 10.2337/db13-0844. PMID 24065795
- [Background] McGill CR, Fulgoni VL 3rd, Devareddy L. Ten-year trends in fiber and whole grain intakes and food sources for the United States population: National Health and Nutrition Examination Survey 2001-2010. Nutrients. 2015 Feb 9;7(2):1119-30. doi: 10.3390/nu7021119. PMID 25671414
- [Background] Sonnenburg ED, Sonnenburg JL. Starving our microbial self: the deleterious consequences of a diet deficient in microbiota-accessible carbohydrates. Cell Metab. 2014 Nov 4;20(5):779-786. doi: 10.1016/j.cmet.2014.07.003. Epub 2014 Aug 21. PMID 25156449